CLINICAL TRIAL: NCT01421485
Title: Integrated Mental Health Treatment & HIV Prevention for Court-Involved Youth
Acronym: ITP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01MH087520-01A2 (NIH)
Record Dates: First submitted 2011-08-19; First posted 2011-08-22 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: HIV Prevention
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrated treatment Program (Experimental)
  Interventions: Behavioral: Integrated treatment program
- Treatment as Usual (Active Comparator)
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Integrated treatment program — CBT, psychopharmacological treatment, family treatment, HIV prevention, case management
  Arms: Integrated treatment Program
Behavioral: Treatment as Usual — Treatment in community, case management
  Arms: Treatment as Usual

SUMMARY:
Youth and young adults in the juvenile justice system have a high prevalence of concurrent psychiatric and substance use disorders and are also at high risk for HIV. However, even when the disorders and risks are recognized, most programs do not address all of these important problems and long-term efficacy for all outcomes simultaneously has yet to be demonstrated for these multi-problem youth. Adverse outcomes for youth include partially treated or relapsing psychiatric disorders, continued substance abuse, unchanged HIV risk, and further legal problems. This project, in collaboration with the Rhode Island Family Court, with whom we have existing collaborations, will address these issues by implementing an Integrated Treatment Program (ITP) that targets mental health/substance abuse disorders and HIV risk. ITP is novel by targeting multiple adolescent problems simultaneously, involving parents to augment change, and its delivery within the Family Court. This study will extend our previous efficacious interventions among youth with psychiatric disorders to court-involved youth. Adolescents and their parents will be enrolled from the Rhode Island Family Court Mental Health Clinic where youth aged 13-17 are referred by judges for comprehensive assessment and referral for treatment. This randomized controlled trial will test the efficacy, among 200 sexually active court-involved youth who need outpatient treatment, of the novel, integrated treatment (ITP, n=100) as compared to enhanced standard care in community outpatient services (ESC, n=100) over an 18-month period (6 months of ITP or ESC and 12 months of follow-up). ITP consists of three components: 1) individual cognitive behavioral therapy which includes a motivational interviewing component and is modular-based to address concurrent mental health and substance abuse issues; 2) family and parent training sessions to address parental communication and monitoring to support risk reduction among youth; 3) multifamily group workshops to address HIV risk, family communication and peer resistance skills. Youth in both conditions (ITP and ESC) will receive similar case management services from the court and psychiatric medication management (if needed) from a study psychiatrist. ITP will be compared to ESC on reductions in sexual risk behavior, substance use, symptoms of psychiatric disorders, and legal offenses.

ELIGIBILITY:
* Adolescents from 13 -17 years of age who report unprotected sex in the past 90 days
* Determined to be in need of mental health treatment by evaluation from the RIFC Mental Health Clinic and so ordered by the judge
* Parent available to participate in the program
* Parent and adolescent English speaking -Adolescent assent and parent/legal guardian consent. -

Exclusion Criteria:

* DSM-IV diagnosis of Obsessive Compulsive Disorder, Pervasive Developmental Disorder, or Schizophrenia as the primary, impairing diagnosis
* IQ less than 70 as determined by the Kaufman Brief Intelligence Test-2 (K-BIT-2)
* Sexual offense charge pending or conviction
* Self-report of HIV infection
* Self-report of current pregnancy
* Wish to remain in mental health and/or medication treatment with an outside provider

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 170 (Actual)
Dates: Start 2011-08; Primary Completion 2015-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Unprotected Sex Acts | Past 90 Days

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Olsen EM, Whiteley LB, Tolou-Shams M, Esposito-Smythers C, Brown LK. Family Factors Associated With Delinquency Outcomes in Court-Involved Youth in Mental Health Treatment. JAACAP Open. 2024 Jul 8;3(3):678-688. doi: 10.1016/j.jaacop.2024.05.004. eCollection 2025 Sep. PMID 40922765